CLINICAL TRIAL: NCT01851343
Title: An Open-Label, Phase 1 Study to Assess the Safety and Tolerability of Bone Marrow Stromal Cell Infusion for the Treatment of Moderate to Severe Inflammatory Bowel Disease
Brief Title: Bone Marrow Stromal Cells for Inflammatory Bowel Diseases
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130077; 13-I-0077
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2017-07-12

CONDITIONS: Inflammatory Bowel Disease
Keywords: Stem Cell Infusion; Crohns; Ulcerative Colitis; Inflammation; Diarrhea
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Inflammation; Diarrhea

ARMS (1):
- 1 (Experimental): All patients will receive the same treatment
  Interventions: Other: Bone Marrow Stromal Cell (BMSC) Infusion

INTERVENTIONS:
Other: Bone Marrow Stromal Cell (BMSC) Infusion — Subjects will receive 4 weekly BMSC infusions and be monitored for AEs as well as for clinical improvement and mucosal healing.

SUMMARY:
Background:

- Bone marrow stromal cells (BMSCs) are cells that can develop into other tissue types, including bone, cartilage, marrow, and blood cells. However, BMSCs are not stem cells there is no evidence that after infusion into another person that BMSCs change into any other cells. Research suggests that BMSCs can travel to different parts of the body and work with immune cells to reduce inflammation and help repair damaged tissues. BMSC infusions have been used in tests to treat moderate to severe inflammatory bowel disease, like Crohn's disease (CD) or ulcerative colitis (UC). These tests have shown some good results, but more research is needed to study their safety and effectiveness. Researchers want to see how well BMSC infusions work to treat CD and UC. The BMSCs will be collected from volunteer donors.

Objectives:

- To look at the safety and effectiveness of BMSC infusions for moderate to severe CD and UC.

Eligibility:

- Individuals between 18 and 65 years old with moderate or severe inflammatory bowel disease (CD or UC) that has not responded to standard treatment.

Design:

* Participants will have two screening visits. The first will be 15 to 30 days before the first BMSC infusion. The second will be within 14 days of the first BMSC infusion.
* At the first screening visit, participants will have a physical exam and medical history. They will provide blood, urine, and stool samples. They will also give information about their symptoms and quality of life.
* At the second screening visit, participants will have their vital signs (like blood pressure and heart rate) measured. They will also provide blood samples, and have a colonoscopy with biopsies.
* During treatment, participants will have one BMSC infusion per week for 4 weeks. Blood and urine samples will be collected at each treatment visit.
* One week after the last infusion, participants will have a study visit. The tests from the first and second screening visits will be repeated.
* There will be six follow-up visits at 1, 2, 3, 6, 12, and 24 months after the last study visit. Participants will repeat the tests from the first screening visit.

DETAILED DESCRIPTION:
Crohn s disease (CD) and ulcerative colitis (UC), the 2 major sub-types of inflammatory bowel disease (IBD), are chronic, life-long conditions characterized by relapsing inflammation of the gastrointestinal tract. CD has a predilection for the small bowel and the proximal large bowel; however, it can affect the gastrointestinal tract discontinuously anywhere. UC mainly affects the distal colon but can involve the entire colon as well. In spite of advances in IBD therapeutics, a significant number of patients continue to have symptoms while on conventional medications. The current protocol proposes to study infusions of allogenic bone marrow stromal cells (BMSCs) for the treatment of active IBD.

The purpose of this study is to evaluate the safety of BMSC infusions in subjects with IBD and to examine the host clinical and immunologic response to BMSCs. BMSCs possess multi-lineage differentiation potential in bone marrow, and aid in the repair of damaged tissue. They suppress the lymphocyte immune response and target sites of inflammation to promote healing through tissue regeneration. Studies are underway examining the utility of BMSCs to treat several conditions including neurologic disorders, myocardial infarctions, rheumatologic disorders, and gastrointestinal disorders including acute graft-versus-host-disease and IBD. Progress in the understanding of the cell populations involved in the pathogenesis of IBD and the discovery of the potential immunologic and regenerative characteristics of BMSCs have created a new potential direction for IBD therapy.

This phase I study will enroll subjects with moderate-to-severe IBD who are refractory to or intolerant of standard therapy. Under the guidance of the NIH Bone Marrow Stromal Cell Transplantation Center, the Cell Processing Section of the Department of Transfusion Medicine at the Clinical Center has developed a procedure for collecting, expanding, and cryopreserving clinical grade BMSCs under an FDA Drug Master File. Marrow will be aspirated from volunteer donors participating on protocol 10-CC-0053 who have passed the standard screening for blood and marrow donors; BMSCs will be expanded in vitro. Since it is not necessary to HLA-match BMSC donors with their recipients, a BMSC repository will be used as the source of BMSCs for this study.

In Arm 1, the safety of the BMSC infusion dosage (4 x 106 cells/kg/dose 10%) and schedule (once a week for 4 weeks) will be evaluated in 3 non-overlapping IBD subjects. Once safety is established in these subjects, subsequent subjects in Arm 2 will be enrolled without overlap restriction. Subjects will return to the clinic for safety and response assessments at 28, 56, 84, and 112 days after the first infusion. Additional safety visits will be performed at 180, 360 and 720 days after the first infusion. Safety will be monitored by a Data and Safety Monitoring Board. Response to study drug will be assessed in all patients by changes in symptom scores, endoscopic/histologic findings, quality of life scores, and immunologic/laboratory parameters. Fifty subjects will be evaluated over a 5-year period.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:

Subjects who meet ALL of the following criteria will be considered for enrollment into this study:

1. Be 18 to 65 years of age, inclusive, as of the date of enrollment.
2. Be willing to take appropriate measures to avoid pregnancy during the study period. Subject to the judgment and discretion of the PI, participants who meet ANY of the criteria listed immediately below, as well as male participants who are in a monogamous relationship with a woman who meets ANY of the criteria below, may not be required to take any pregnancy avoidance measures (e.g. barrier methods). Such participants will be counseled on risks at the time of consent and at appropriate points (e.g. when pregnancy testing occurs) during the study:

   1. Females who have had their uterus, and/or BOTH ovaries removed
   2. Females who have had BOTH fallopian tubes surgically tied or removed
   3. Females who have undergone other permanent birth control procedures, such as endometrial ablation or sterilization (such as Essure or Novasure), and have had any required follow up testing to confirm the effectiveness of the permanent birth control procedure.
   4. Females who are above the age of 50 and have spontaneously had no menses at any point during the past 12 or more consecutive months (i.e. have reached menopause).
   5. Females who, in the conservative and reasonable judgment of the PI (e.g. due to sexual orientation, or serious life choice), from the time of enrollment until

      12 weeks after the last BMSC infusion, will NOT participate in any potentially reproductive sexual contact (i.e. sexual intercourse with a male partner).
   6. Males who have had a vasectomy and have had the follow-up testing confirming zero sperm count in their semen.
3. Any subject who does NOT meet the criteria listed in #2 above, will be appropriately counseled on reproductive risks and pregnancy avoidance, and will be required to adhere to the following measures, as agreed upon by the subject and the PI until at least 12 weeks after the last BMSC infusion:

   1. A highly effective hormonal method to prevent pregnancy [e.g. CONSISTENT, CONTINUOUS use of contraceptive pill, patch, ring, implant or injection], and/or IUD or equivalent.

      IN ADDITION TO
   2. A barrier method to be used at the time of potentially reproductive sexual activity (e.g. [male/female condom, cap, or diaphragm] + spermicide).
   3. Male participants will be appropriately counseled on risks and must agree to consistently use effective contraception with female sexual partners through the Day 112 study visit to avoid a pregnancy that could be affected by the study drug. Appropriate measures to avoid pregnancy and trial related risks in sexual partners, per the PI s judgment, must be agreed to and practiced.

   NOTE: Most of the above interventions to prevent pregnancy must be implemented at a particular time in the menstrual cycle, and may not be immediately effective. Trial activity that may pose a reproductive risk may NOT occur until the above contraceptive measures are fully effective and must continue until at least 12 weeks after the last BMSC infusion.
4. Have a diagnosis of CD or UC that has been endoscopically or radiographically confirmed at least 6 months prior to screening.
5. Have either active CD symptoms as defined by a CDAI score between 220 and 450, inclusive, as measured for 7 consecutive days during screening, or active UC as defined by a SCCAI score greater than or equal to 6.
6. The patient must have demonstrated an inadequate response to, loss of response to, or intolerance of at least 1 of the following agents as defined below:

   * Corticosteroids

     * Signs and symptoms of persistently active disease despite a history of at least one 4-week induction regimen that included a dose equivalent to prednisone 30 mg daily orally for 2 weeks or intravenously for 1 week OR
     * Two failed attempts to taper corticosteroids to below a dose equivalent to prednisone 10 mg daily orally on 2 separate occasions OR
     * History of intolerance of corticosteroids (including, but not limited to Cushing s syndrome, osteopenia/osteoporosis, hyperglycemia, insomnia, infection)
   * Immunomodulators

     * Signs and symptoms of persistently active disease despite a history of at least one 8 week regimen of oral azathioprine (greater than or equal to 1.5 mg/kg) or 6-mercaptopurine mg/kg (greater than or equal to 0.75 mg/kg) OR
     * Signs and symptoms of persistently active disease despite a history of at least one 8 week regimen of methotrexate (greater than or equal to 12.5 mg/week) OR
     * History of intolerance of at least one immunomodulator (including, but not limited to nausea/vomiting, abdominal pain, pancreatitis, LFT abnormalities, lymphopenia, TPMT genetic mutation, infection)
   * TNF alpha antagonists

     * Signs and symptoms of persistently active disease despite a history of at least one 4 week induction regimen of 1 of the following agents

       * Infliximab: 5 mg/kg IV, 2 doses at least 2 weeks apart
       * Adalimumab: one 80 mg SC dose followed by one 40 mg dose at least 2 weeks apart
       * Certolizumab pegol: 400 mg SC, 2 doses at least 2 weeks apart OR
     * Recurrence of symptoms during scheduled maintenance dosing following prior clinical benefit (discontinuation despite clinical benefit does not qualify) OR
     * History of intolerance of at least 1 TNF antagonist (including, but not limited to infusion-related reaction, demyelination, congestive heart failure, infection)
7. May be receiving a therapeutic dose of the following drugs:

   * Oral 5-ASA compounds provided that the dose has been stable for the 2 weeks immediately prior to enrollment
   * Oral corticosteroid therapy (prednisone at a stable dose less than or equal to 30 mg/day, budesonide at a stable dose less than or equal to 9 mg/day, or equivalent steroid) provided that the dose has been stable for the 4 weeks immediately prior to enrollment if corticosteroids have just been initiated, or for the 2 weeks immediately prior to enrollment if corticosteroids are being tapered
   * Probiotics (e.g., Culturelle, Saccharomyces boulardii) provided that the dose has been stable for the 2 weeks immediately prior to enrollment
   * Antidiarrheals (e.g., loperamide, diphenoxylate with atropine) for control of chronic diarrhea
   * Azathioprine or 6-mercaptopurine provided that the dose has been stable for the 8 weeks immediately prior to enrollment
   * Methotrexate provided that the dose has been stable for the 8 weeks immediately prior to enrollment
   * Antibiotics used for the treatment of CD (i.e., ciprofloxacin, metronidazole) provided that the dose has been stable for the 2 weeks immediately prior to enrollment
8. Subjects must agree to have samples of their blood and tissue samples stored for potential future research use.
9. Be willing to take appropriate measures to avoid pregnancy until at least 12 weeks after the last BMSC infusion. All subjects will be informed of the potential risks of BMSC during pregnancy and counseled on pregnancy avoidance appropriate to the subject s circumstances (e.g. fertility status, medical contraindications to hormonal birth control, and/or personal or religious beliefs regarding pregnancy avoidance). Subject to thejudgement and discretion of the PI, some subjects may not need to take pregnancy avoidance measures.
10. Subjects must have a primary medical care provider.

SUBJECT EXCLUSION CRITERIA

Subjects who meet ANY of the following criteria will be excluded from participation in this study:

1. Subjects who are currently taking greater than or equal to 20 mg of prednisone per day. Subjects on corticosteroids must be on a stable dose for at least 4 weeks.
2. Concomitant treatment with anti-TNF therapy (or other biological therapy) or with Entyvio/vedolizumab. The following washout period will be required for subjects to be eligible to participate in the trial:

   1. Three months washout prior to baseline for certolizumab or natalizumab.
   2. Two months washout prior to baseline for adalimumab, etanercept, infliximab, and Entyvio/vedolizumab.
   3. One month washout prior to baseline for cyclosporine, mycophenolate,

   pimecrolimus, tacrolimus, and any other systemic immunosuppressants.
3. Pregnant or breastfeeding. Serum pregnancy test must be negative at screening for female subjects of childbearing potential. Urine pregnancy test must remain negative at each of the four infusion visits.
4. Subject does not agree to pregnancy avoidance measures required to prevent pregnancy during participation in the study, or meet criteria that would exempt them from contraceptive measures.
5. Has clinically significant systemic infection (e.g., chronic or acute infection, urinary tract infection, upper respiratory tract infection) within one month of screening and no opportunistic infection within six months of screening. Has a history or presence of recurrent or chronic infection (e.g. viral infections [including hepatitis B or C, HIV], bacterial infections, systemic fungal infections, or syphilis).
6. Has a positive Quantiferon-TB Gold (QFT-G) test, indicating tuberculosis infection, at time of screening. A QFT-G will not be done in a subject who has received tuberculosis vaccination; these subjects will be eligible to participate if latent tuberculosis can be excluded with a chest x-ray (CXR).
7. Received an agent not approved by the FDA for marketed use in any indication or any small molecule inhibitors (e.g., Naltrexone) within 90 days of beginning the screening CDAI diary or at any time during the screening window. This includes medications used to treat IBD as an off-label use (at the discretion of the investigator).
8. Has abnormal hematological and biochemical parameters, including:

   * Neutrophil count <1500 cells/mm(3).
   * Hemoglobin <9 g/dL.
   * Platelet count less than or equal to150,000 cells/mm(3).
   * Creatinine greater than or equal to1.2 times the upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) greater than or equal to2 times ULN.
   * Prothrombin time-International Normalized Ratio (PT-INR) >2 and/or on chronic anticoagulation medications.
   * If total bilirubin is greater than 1.2 mg/dL, then direct bilirubin can be no more than 70% of the total, up to a direct bilirubin of 2.0 mg/dL.
9. Has active infection with enteric pathogens as evidenced by positive microbiological culture of stool.
10. Has active cytomegalovirus (CMV) infection. CMV polymerase chain reaction (PCR) testing will be performed on biopsies taken during the time of initial colonoscopy in order to exclude CMV.
11. Has a history of low-grade or high-grade colonic mucosal dysplasia.
12. Has a history of uveitis or iritis within the previous two months. This is due to the concern that BMSCs may home to sites of active inflammation.
13. Had bowel surgery other than perianal (e.g., fistulotomy, seton placement, abscess drainage) within 6 months prior to beginning the CDAI screening diary or drawing screening blood samples.
14. Has surgical changes to gut anatomy that preclude administration of clinical activity indicies including but not limited to ileostomy, colostomy, or subtotal colectomy with ileorectal anastomosis.
15. Has known or suspected short bowel syndrome.
16. Requires parenteral or total parenteral nutrition.
17. Has a history of cancer, other than non-melanomatous cancer of the skin, within the past 5 years.
18. Unwillingness or inability to comply with study requirements.
19. Has any medical or psychiatric condition that, in the opinion of the investigator, contraindicates participation in this protocol.
20. Has only small bowel IBD that is inaccessible by standard colonoscopy to obtain research biopsies. For this reason patients with only upper gastrointestinal IBD are also excluded.
21. Refuses to abstain from using COX-2 inhibitors or NSAIDs throughout the 4 week study drug infusion period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01-27; Primary Completion 2017-07-12 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as measured by the presence of any AEs | Day 0 through Week 16

SECONDARY OUTCOMES:
Proportion of subjects who achieve clinical response and remission, mucosal healing, change in immunologic parameters and stability of remission/response at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ivan J Fuss, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Devine SM, Cobbs C, Jennings M, Bartholomew A, Hoffman R. Mesenchymal stem cells distribute to a wide range of tissues following systemic infusion into nonhuman primates. Blood. 2003 Apr 15;101(8):2999-3001. doi: 10.1182/blood-2002-06-1830. Epub 2002 Dec 12. PMID 12480709
- [Background] Nauta AJ, Fibbe WE. Immunomodulatory properties of mesenchymal stromal cells. Blood. 2007 Nov 15;110(10):3499-506. doi: 10.1182/blood-2007-02-069716. Epub 2007 Jul 30. PMID 17664353
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814